CLINICAL TRIAL: NCT01752283
Title: Combination of Video-assisted Thyroid Surgery and Hypnosis as a Complete Minimally Invasive Approach: a Comparative Pilot Study
Brief Title: Video-assisted Thyroid Surgery and Hypnosis in Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Mourad, MD, PhD, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Video-Hypnose
Record Dates: First submitted 2012-10-31; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Surgery
Keywords: Videoassited; Thyroidectomy; Minimal invasive surgery; General anesthesia; Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypnosis and local anesthesia (Experimental): video-assisted thyroidectomy under hypnosis and local anesthesia.
  Interventions: Procedure: video-assisted thyroidectomy
- General anesthesia (Active Comparator): Video-assisted thyroidectomy under general anesthesia
  Interventions: Procedure: video-assisted thyroidectomy

INTERVENTIONS:
Procedure: video-assisted thyroidectomy — Experimental arm: video-assisted thyroidectomy under local anesthesia and hypnosis
Procedure: Video-assisted thyroidectomy — video-assisted thyroidectomy under general anesthesia

SUMMARY:
The study is aimed to investigate the safety and feasibility of Video-assisted thyroidectomy under hypnosis in comparison to general anesthesia

DETAILED DESCRIPTION:
Summary of the project

video-assisted thyroidectomy (MIVAT): General anesthesia (GA) versus hypnosis (HY)

Investigators

Prof. Michel Mourad*, Dr. Christine Watremez **, Prof. Fabienne Roelants**

* Surgery and Abdominal Transplantation Division

** Department of Anesthesiology,

Université Catholique de Louvain, Cliniques Universitaires Saint-Luc, Avenue Hippocrate 10, 1200 Brussels, Belgium

1. Aim

   The aim of this pilot study is to prospectively investigate, in a consecutive series of patients, the feasibility and safety of MIVAT under HY associated with local anesthesia, compared to GA.
2. Inclusion criteria

   * Adult patients candidates to total or partial thyroidectomy.
   * ASA 1, 2 or 3
   * One surgeon (MM)
   * Informed consent
3. Exclusion criteria

   * Age <18 years
   * The presence of familial medullary thyroid cancers
   * Suspicious or metastatic lymph nodes
   * Redo surgery
   * ASA 4 patients
   * Patients with chronic pain
   * Deaf people
   * Patients with psychiatric diseases
   * Known recurrent nerve paralysis
4. Outcome evaluation

   * Primary outcomes: safety and feasibility.
   * During surgery, considered events for analysis should include operating time (from skin incision to skin closure), total time in the operating room, intraoperative bleeding, drug consumption, Hemodynamic changes and conversion rates from MIVAT to a conventional approach and from HY to GA.
   * After surgery, comparative variables for analysis should include: drug consumption, hospital stay, calcemia, and vocal cord abnormality on the basis of day-one laryngoscopy performed by an ENT doctor not involved in the study.
5. Patients selection and study groups:

Selection of patients for MIVAT is based on the size of the gland and nodules, provided that the craniocaudal axis of the lobes did not exceed 7cm and the largest transversal diameter was less than 3.5cm. All patients who are assigned to undergo MIVAT are instructed about the possibility of conversion to a conventional approach. The patients are left free to choose the type of anesthesia they prefere for their surgical intervention. They have to give informed consent before the procedure.

A. General anesthesia group:

Premedication:

* Lorazepam 0.5 mg 1 h before surgery
* ECG, NIBP, SaO2
* VVP + NaCl 0.9 % 500 mL + taradyl 0.5 mg / kg (<30 mg)

Induction:

* Remifentanil 0.05 µg/kg/min
* Propofol 2 mg/kg
* Intubation with an armored endotracheal tube specially devised for neuromonitoring of the vocal cords.

During surgery:

* Sevoflurane / Remifentanil

B. Hypnosis group:

Premedication:

* Lorazepam 0.5 mg 1 h avant l'intervention
* ECG, NIBP, SaO2
* VVP + NaCl 0.9 % 500 mL + taradyl 0.5 mg / kg (< 30 mg)

Induction and during surgery:

* Remifentanil modified as requested
* Induction of hypnosis according to Milton Eriksson technique
* Midazolam (titrated 0.1 mg/0.1mg) if needed as anxiolytic.
* Local anesthesia mixture (lidocaine 0.5%/ropivacaine 0.25%) to be administered by the surgeon along the incision line 5 minutes before making the skin incision.

ELIGIBILITY:
Inclusion Criteria:

* The selection of patients for MIVAT was achieved according to the size of the gland and nodules provided that the cranio-caudal axis of the lobes does not exceed 7 centimeters and the largest transversal diameter is less than 3.5 centimeters
* Age >18 years

Exclusion Criteria:

* No previous neck surgery
* No known malignancy
* No history of neck irradiation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Feasibility | Intraoperative
  To assess technical feasibility

SECONDARY OUTCOMES:
Operating time | during surgery
Intraoperative bleeding | During surgery
Conversion to general anesthesia | During surgery
Conversion from video-assisted technique to conventional surgery | During surgery

OTHER OUTCOMES:
Hemodynamic changes | During surgery
Drug consumption | During surgery and up to 6 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michel Mourad, MD, PhD, Principal Investigator — Cliniques Universitaires Saint-Luc. 10 Avenue Hippocrate, 10. 1200 Bruxelles
Locations (1):
- Cliniques Universitaires Saint-Luc. 10 Avenue Hippocrate, Brussels, Belgium